CLINICAL TRIAL: NCT03573739
Title: Impact of Early Low-Calorie Low-Protein Versus Standard-Calorie Standard-Protein Feeding on Outcomes of Ventilated Adults With Shock: a Randomised, Controlled, Multicentre, Open-label, Parallel-group Study (NUTRIREA-3)
Brief Title: Impact of Early Low-Calorie Low-Protein Versus Standard Feeding on Outcomes of Ventilated Adults With Shock
Acronym: NUTRIREA3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC18_0006
Record Dates: First submitted 2018-06-07; First posted 2018-06-29 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Critical Illness; Shock; Mechanical Ventilation; Critical Illness Myopathy; Nosocomial Infection
MeSH Terms: conditions — Critical Illness; Shock; Cross Infection

STUDY DESIGN:
Intervention Model Description: This multicentre randomised controlled open trial compares two parallel groups of patients receiving mechanical ventilation and vasoactive amine therapy and given early nutritional support according to one of two strategies: early calorie/protein restriction (6 kcal/kg/d/0.2-0.4 g/kg/d: Low group) or standard calorie/protein targets (25 kcal/kg/d/1.0-1.3g/kg/d: Standard group) at the acute phase of ICU management (D0-D7).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low group (Experimental): Patients randomized in the "low group" will receive a low-calorie low-protein nutrition regimen during the acute phase.
  Interventions: Procedure: low-calorie low-protein
- Standard group (Active Comparator): Patients randomized in the "standard group" will receive a standard-calorie/standard-protein nutrition regimen during the acute phase.
  Interventions: Procedure: standard-calorie/standard-protein

INTERVENTIONS:
Procedure: low-calorie low-protein — In the low-calorie low-protein (Low) group, the calorie target will be 6 kcal/kg/day and the protein target 0.2-0.4 g/kg/d during the acute phase, i.e. from D0 to D7. On D8, the calorie target will be 30 kcal/kg/d and the protein target 1.2-2.0 g/kg/d.
  Arms: Low group
Procedure: standard-calorie/standard-protein — In the standard-calorie/standard-protein (Standard) group, the first-line calorie target calculated based on body weight is 25 kcal/kg/day and the protein target 1.0-1.3 g/kg/d during the acute phase, i.e. from D0 to D7. On D8, the calorie target will be 30 kcal/kg/d and the protein target 1.2-2.0 g/kg/d.
  Arms: Standard group

SUMMARY:
Among critically ill patients requiring mechanical ventilation and catecholamines for shock, nearly 40% to 50% die, and functional recovery is often delayed in survivors. International guidelines include early nutritional support (≤48 h after admission), 20-25 kcal/kg/d at the acute phase, and 1.2-2 g/kg/d protein. These targets are rarely achieved in patients with severe critically illnesses. Recent data challenge the wisdom of providing standard amounts of calories and protein during the acute phase of critical illness. Studies designed to improve enteral nutrition delivery showed no outcome benefits with higher intakes. Instead, adding parenteral nutrition to increase intakes was associated with longer ICU stays and more infectious complications. Studies suggest that higher protein intakes during the acute phase may be associated with greater muscle wasting and ICU-acquired weakness. The optimal calorie and protein supply at the acute phase of severe critical illness remains unknown. NUTRIREA-3 will be the first trial to compare standard calorie and protein feeding complying with guidelines to low-calorie low-protein feeding potentially associated with improved muscle preservation, translating into shorter mechanical ventilation and ICU-stay durations, lower ICU-acquired infection rates, lower mortality, and better long-term clinical outcomes. This multicentre, randomized, controlled, open trial will compare, in patients receiving mechanical ventilation and treated with vasoactive agent for shock two strategies for initiating nutritional support at the acute phase of ICU management (D0-D7): early calorie/protein restriction (6 kcal/kg/d/0.2-0.4 g/kg/d, Low group) or standard calorie/protein targets (25 kcal/kg/d/1.0-1.3 g/kg/d, Standard group). Patients in both groups will receive enteral or parenteral nutrition appropriate for their critical illness. Two alternative primary end-points will be evaluated: all-cause mortality by day 90 and time to discharge alive from the ICU. Second end-points will be calories and proteins delivered, nosocomial infections, gastro-intestinal complications, glucose control, liver dysfunctions, muscle function at the time of readiness for ICU discharge and quality of life at 3 months and 1 year after study inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation started in the ICU within the past 24 h, or started before ICU admission with ICU admission within the past 24 h, for an expected duration of at least 48 hours after inclusion
* Treatment with a vasoactive agent for shock (adrenaline, dobutamine, or noradrenaline)
* Nutritional support expected to be started within 24 h after intubation or within 24 h after ICU admission when mechanical ventilation was started before ICU admission
* Age older than 18 years
* Patient and/or next-of-kin informed about the study and having consented to participation in the study. If the patient is unable to receive information and no next-of-kin can be contacted during screening for the study, trial inclusion will be completed as an emergency procedure by the ICU physician, in compliance with the French law.

Exclusion Criteria:

* Specific nutritional needs, such as pre-existing long-term home enteral or parenteral nutrition, for chronic bowel disease
* Dying patient, not-to-be-resuscitated order, or other treatment limitation decision at ICU admission
* Pregnancy, recent delivery, or lactation
* Adult under guardianship
* Department of corrections inmate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3044 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Time to discharge alive from the ICU. | From date of ICU admission until the date of first documented date when predefined clinical conditions for ICU discharge are fulfilled, an average of 10 days.
  A patient will be considered ready for ICU discharge by the bedside physicians as soon as all predefined clinical conditions for ICU discharge are fulfilled, regardless of ward-bed availability.
D-90 mortality | 90 days
  All-cause mortality by day 90

SECONDARY OUTCOMES:
Number of calories (in kcal) delivered daily enterally and/or parenterally | from day 0 to day 7
Ratio of prescribed over calories delivered | from day 0 to day 7
  Ratio (as a %) of prescribed over calories delivered daily enterally and/or parenterally
Proportion of patients who achieved their calorie target | from day 0 to day 7
  Proportion of patients who achieved their calorie target
Protein supply | from day 0 to day 7
  Protein supply (g) given daily enterally and/or parenterally
Volume of fluids | from day 0 to day 7
  Volume of fluids (in mL) received daily
Changes in Sequential Organ Failure Assessment (SOFA) score | from day 0 to day 7
  SOFA scores can range from 0 (no organ failure) to 24 (most severe level of multi-organ failure).
Changes in daily maximum blood glucose levels | from day 0 to day 7
Proportion of patients with hypoglycaemia | from day 0 to day 7
insulin dose | from day 0 to day 7
  Total insulin dose received daily
insulin treatment | from day 0 to readiness for ICU discharge, an average of 10 days
  Days on insulin treatment
Proportion of patients with at least one ICU-acquired infection. | from day 0 to readiness for ICU discharge, an average of 10 days
Proportion of patients with each type ICU-acquired infection | from day 0 to readiness for ICU discharge, an average of 10 days
  e.g. (Ventilator-associated pneumonia, bacteremia, Central venous catheter-related infections, Urinary tract infections, soft tissue infections).
Proportion of patients with at least one episode of vomiting or regurgitation while on mechanical ventilation | from day 0 to extubation, an average of 7 days
Proportion of patients with at least one episode of liver dysfunction during follow-up | from day 0 to readiness for ICU discharge, an average of 10 days
Proportion of patients with at least one episode of diarrhoea | from day 0 to extubation, an average of 7 days
  defined as liquid stools in a volume greater than 300 mL/24 hours in patients with a faecal collector or as more than four loose stools/24 hours
Proportion of patients with at least one episode of constipation | from day 0 to extubation, an average of 7 days
  no stool for more than 6 days
Proportion of patients with at least one documented episode of bowel ischaemia | from day 0 to readiness for ICU discharge, an average of 10 days
Mean changes in serum albumin | from day 0 to day 7 and readiness for ICU discharge, an average of 10 days
  measured at baseline, at the end of mechanical ventilation, on day 7 (in patients on mechanical ventilation for more than 7 days), and at ICU discharge
Mean changes in serum pre-albumin | from day 0 to day 7 and readiness for ICU discharge, an average of 10 days
  measured at baseline, at the end of mechanical ventilation, on day 7 (in patients on mechanical ventilation for more than 7 days), and at ICU discharge
Changes in serum C-reactive protein (CRP) | from day 0 to day 7 and readiness for ICU discharge, an average of 10 days
  measured at baseline, at the end of mechanical ventilation, on day 7 (in patients on mechanical ventilation for more than 7 days), and at ICU discharge
Changes in mean body weight | from day 0 to day 7 and readiness for ICU discharge, an average of 10 days
  determined at baseline, on day 7, and at ICU discharge
Hospital stay | from day 0 to hospital discharge, an average of 23 days
  Hospital stay length (days in hospital)
Duration of mechanical ventilation | from day 0 to extubation, an average of 7 days
  Days on mechanical ventilation
ICU mortality | from day 0 to ICU discharge, an average of 23 days
  Proportions of patients dead during the ICU stay
Mortality at day 28 | from day 0 to day 28
  Proportions of patients dead until day 28 after randomization
Hospital mortality | from day 0 to hospital discharge, an average of 23 days
  Proportions of patients dead during the hospital stay
Proportions of patients mobilized | from day 0 to day 7
  Evaluation of mobilisation during the ICU stay using predetermined criteria.
Total number of active mobilizations | from day 0 to day 7
  Evaluation of mobilisation during the ICU stay using predetermined criteria.
Muscle function | On the day of readiness for ICU discharge, an average of 10 days
  Muscle function at the time of readiness for ICU discharge as assessed with the Medical Research Council (MRC) score. The MRC score ranges from 0 (no muscle activity) to 60 (normal muscle function).
Proportion of patients with at least one criterion for persistent altered health status | On the day of readiness for ICU discharge, an average of 10 days
  at the time of readiness for ICU discharge
SF-36 score | 3 months and 1 year after study inclusion
  The Short Form (SF)-36 is a multipurpose health survey with 36 questions. Questionnaires will be completed during a phone call to the patient by an independent blinded research nurse or psychologist.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Reignier, MD, PhD, Principal Investigator — Nantes University Hospital
Locations (59):
- France (58):
  - Chu de La Reunion Site Nord, Saint-Denis, La Réunion
  - Chu Amiens Picardie, Amiens
  - CHU Angers, Angers
  - Centre Hospitalier D'Angouleme, Angoulême
  - Ch Annecy-Genevois, Annecy
  - Centre Hospitalier D'Argenteuil, Argenteuil
  - Hôpital du bois brulé, Beauvais
  - Hôpital Nord Franche Comté, Belfort
  - Chu Jean Minjoz, Besançon
  - Hôpital de Béthune, Béthune
  - Hôpital Avicenne AP-HP, Bobigny
  - Hopital Pellegrin Chu, Bordeaux
  - CHU Cavale Blanche, Brest
  - Ch Chartres Louis Pasteur, Chartres
  - Chu Gabriel Montpied, Clermont-Ferrand
  - Hopital Louis Mourier (Ap-Hp), Colombes
  - Ch Dieppe, Dieppe
  - Chu Bocage, Dijon
  - Hôpital Raymond-Poincaré, Garches
  - Hôpital Michalon, Grenoble
  - Chd Les Oudairies, La Roche-sur-Yon
  - Chu Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Du Mans, Le Mans
  - CH Emile Roux, Le Puy-en-Velay
  - Centre Hospitalier de Lens, Lens
  - Chr - Hopital Roger Salengro, Lille
  - CH Saint-Philibert, Lomme
  - Hopital de La Croix-Rousse, Lyon
  - Hopital Edouard Herriot, Lyon
  - Centre Hospitalier Marc Jacquet, Melun
  - Centre Hospitalier de Montauban, Montauban
  - Hopital Saint Eloi, Montpellier
  - Ctre Hosp Intercomm Andre Gregoire, Montreuil
  - Chu de Nantes, Nantes
  - CHU Nantes, Nantes
  - Chr D'Orleans, Orléans
  - Hopital Lariboisiere, Paris
  - Hôpital Saint Louis (AP-HP), Paris
  - Hopital Saint Antoine, Paris
  - Hopital Pitie Salpetriere, Paris
  - CHU Paris Cochin, Paris
  - G.I.H. Bichat / Claude Bernard (Ap-Hp), Paris
  - Hopital Europeen Georges Pompidou, Paris
  - CH Pau, Pau
  - Chu La Miletrie, Poitiers
  - C.H.R. Pontchaillou, Rennes
  - C.H. de Rodez Hopital Jacques Puel, Rodez
  - Hopital Charles Nicolle Chu Rouen, Rouen
  - CH Saint Brieuc, Saint-Brieuc
  - Ch General Delafontaine, Saint-Denis
  - CHU de Saint Etienne, Saint-Priest-en-Jarez
  - Hopital Broussais, St-Malo
  - Hôpital de Hautepierre CHU de Strasbourg, Strasbourg
  - Hopital Foch, Suresnes
  - CH de Bigorre, Tarbes
  - CHU DE TOURS Bretonneau, Tours
  - CH Valenciennes, Valenciennes
  - Centre Hospitalier Bretagne Atlantique - Vannes Auray, Vannes
- CHU Pointe à Pitre - Abymes, Pointe-à-Pitre, Guadeloupe

REFERENCES:
- [Derived] Reignier J, Plantefeve G, Mira JP, Argaud L, Asfar P, Aissaoui N, Badie J, Botoc NV, Brisard L, Bui HN, Chatellier D, Chauvelot L, Combes A, Cracco C, Darmon M, Das V, Debarre M, Delbove A, Devaquet J, Dumont LM, Gontier O, Groyer S, Guerin L, Guidet B, Hourmant Y, Jaber S, Lambiotte F, Leroy C, Letocart P, Madeux B, Maizel J, Martinet O, Martino F, Maxime V, Mercier E, Nay MA, Nseir S, Oziel J, Picard W, Piton G, Quenot JP, Reizine F, Renault A, Richecoeur J, Rigaud JP, Schneider F, Silva D, Sirodot M, Souweine B, Tamion F, Terzi N, Thevenin D, Thiery G, Thieulot-Rolin N, Timsit JF, Tinturier F, Tirot P, Vanderlinden T, Vinatier I, Vinsonneau C, Voicu S, Lascarrou JB, Le Gouge A; NUTRIREA-3 Trial Investigators; Clinical Research in Intensive Care; Sepsis (CRICS-TRIGGERSEP)Group. Low versus standard calorie and protein feeding in ventilated adults with shock: a randomised, controlled, multicentre, open-label, parallel-group trial (NUTRIREA-3). Lancet Respir Med. 2023 Jul;11(7):602-612. doi: 10.1016/S2213-2600(23)00092-9. Epub 2023 Mar 20. PMID 36958363
- [Derived] Reignier J, Le Gouge A, Lascarrou JB, Annane D, Argaud L, Hourmant Y, Asfar P, Badie J, Nay MA, Botoc NV, Brisard L, Bui HN, Chatellier D, Chauvelot L, Combes A, Cracco C, Darmon M, Das V, Debarre M, Delbove A, Devaquet J, Voicu S, Aissaoui-Balanant N, Dumont LM, Oziel J, Gontier O, Groyer S, Guidet B, Jaber S, Lambiotte F, Leroy C, Letocart P, Madeux B, Maizel J, Martinet O, Martino F, Mercier E, Mira JP, Nseir S, Picard W, Piton G, Plantefeve G, Quenot JP, Renault A, Guerin L, Richecoeur J, Rigaud JP, Schneider F, Silva D, Sirodot M, Souweine B, Reizine F, Tamion F, Terzi N, Thevenin D, Thiery G, Thieulot-Rolin N, Timsit JF, Tinturier F, Tirot P, Vanderlinden T, Vinatier I, Vinsonneau C, Maugars D, Giraudeau B. Impact of early low-calorie low-protein versus standard-calorie standard-protein feeding on outcomes of ventilated adults with shock: design and conduct of a randomised, controlled, multicentre, open-label, parallel-group trial (NUTRIREA-3). BMJ Open. 2021 May 11;11(5):e045041. doi: 10.1136/bmjopen-2020-045041. PMID 33980526